CLINICAL TRIAL: NCT07377422
Title: Safety and Efficacy of a Novel Composite-Tip Guiding Catheter in Transcarotid Artery Stenting Via Transradial Access: A Prospective, Multicenter, Randomized Controlled Trial
Brief Title: Safety and Efficacy of a Novel Composite-Tip Guiding Catheter in Transcarotid Artery Stenting Via Transradial Access
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Guo Xu, Associate Chief Physician, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BC-CR202501; 2025AZC2008 (Other Grant/Funding Number: Beijing Anzhen Hospital. Capital Medical University)
Record Dates: First submitted 2025-12-15; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Transradial Carotid Artery Stenting; Novel Composite-tip Guiding Catheter

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Composite-Tip Transradial Neurovascular Distal Access Catheter (Experimental)
  Interventions: Device: Composite-Tip Transradial Neurovascular Distal Access Catheter
- Straight or Single-Curve Tip Guiding Catheter (Active Comparator)
  Interventions: Device: Straight or Single-Curve Tip Guiding Catheter

INTERVENTIONS:
Device: Composite-Tip Transradial Neurovascular Distal Access Catheter — Carotid Artery Stenting via Transradial Access Using a Composite-Tip Neurovascular Distal Access Catheter
  Arms: Composite-Tip Transradial Neurovascular Distal Access Catheter
Device: Straight or Single-Curve Tip Guiding Catheter — Carotid Artery Stenting via Transradial Access Using Straight or Single-Curve Tip Guiding Catheter
  Arms: Straight or Single-Curve Tip Guiding Catheter

SUMMARY:
This study aims to evaluate the safety and efficacy of the novel composite-tip guiding catheter for transradial access in Carotid Artery Stenting procedures

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Patients who are candidates for endovascular intervention with CTA-confirmed stenosis in the common carotid artery or C1 segment of internal carotid artery(Symptomatic: ≥50% stenosis; Asymptomatic: 70%-99% stenosis）（NASCET criteria) ;

   * Symptomatic carotid artery stenosis: Non-disabling ischemic stroke or transient ischemic symptoms (TIA, including hemispheric events or transient monocular blindness) within 180 days prior to randomization;

     * Asymptomatic Carotid Stenosis: No history or examination findings suggestive of ipsilateral carotid ischemic symptoms(Non-carotid symptoms, contralateral carotid symptoms, symptom onset >180 days prior to randomization, or vertebrobasilar symptoms are classified as asymptomatic).
3. Palpable radial pulse and negative Allen's test (confirming adequate ulnar collateral circulation);
4. Feasible transradial access with achievable device delivery to the target lesion per operator assessment;
5. Patients or legally authorized representatives comprehend the study purpose, voluntarily participate with signed informed consent, and commit to complete follow-up.

Exclusion Criteria:

1. Patients with severe vascular tortuosity/dissection, extensive or diffuse atherosclerotic lesions involving the aortic arch or proximal common carotid artery, or post-surgical anatomy impeding catheter delivery;
2. Severe stenosis, aneurysms ≥5mm in maximum diameter, arteriovenous malformations (AVM), or other significant cerebrovascular diseases in ipsilateral intracranial/extracranial arteries beyond the target vessel;
3. Patients requiring simultaneous bilateral carotid interventions;
4. Contraindicated in patients with severe allergies to interventional devices or agents related to carotid stenting (e.g., lidocaine, contrast agents, aspirin, clopidogrel);
5. Preprocedural mRS ≥3;
6. Progressive stroke within 2 weeks, hemorrhagic transformation of ischemic stroke within 3 months, or spontaneous intracranial hemorrhage within 12 months;
7. Severe hematologic disorders (active bleeding, severe anemia, coagulopathy, or transfusion dependency), severe heart failure, severe hepatic/renal impairment, or acute coronary syndrome;
8. Malignancy or life expectancy <1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2026-01-19 (Estimated); Primary Completion 2027-06-16 (Estimated); Study Completion 2027-08-16 (Estimated)

PRIMARY OUTCOMES:
Transradial Access Success Rate Within 10 Minutes | Intra-procedure

SECONDARY OUTCOMES:
Success Rate of Transradial Access Carotid Artery Stenting | Immediately post-procedure
Primary Success Rate of Transradial Access Establishment | Intra-procedure
Transradial-to-Transfemoral Conversion Rate | Intra-procedure
X-ray Radiation Exposure | Intra-procedure
Clinician User Experience Assessment | Immediately post-procedure
National Institutes of Health Stroke Scale (NIHSS) Score | Pre-discharge
Post-Procedure Modified Rankin Scale (mRS) Score | Pre-discharge
Incidence Rate of Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) | Pre-discharge，30 days post-procedure
Incidence Rate of All-Cause Death | Pre-discharge，30 days post-procedure
Incidence Rate of Any Stroke | Pre-discharge，30 days post-procedure
Incidence Rate of Target Vessel-Related Ischemic Stroke | Pre-discharge，30 days post-procedure
Incidence Rate of Any Myocardial Infarction | Pre-discharge，30 days post-procedure
Incidence Rate of Any Revascularization | Pre-discharge，30 days post-procedure
Incidence Rate of Radial Artery Occlusion | Pre-discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital. Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided